CLINICAL TRIAL: NCT05873439
Title: A Feasibility Study of Genomically Guided Radiation Dose Personalization in the Management of Locally Advanced Non-Small Cell Lung Cancer
Brief Title: Genomically Guided Radiation Dose Personalization in Locally Advanced NSCLC
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MCC 21525
Record Dates: First submitted 2023-05-12; First posted 2023-05-24 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Nonsmall Cell Lung Cancer; Nonsmall Cell Lung Cancer, Stage II; Nonsmall Cell Lung Cancer Stage III; Unresectable Non-Small Cell Lung Carcinoma
Keywords: Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Arm A: RSI predicts dose ≤ 60 Gy (Experimental): Participants will receive standard RT dose of 60Gy in 30 fractions targeting the primary tumor and any involved regional lymph nodes.
  Interventions: Radiation: Genomically Guided Radiation Therapy (RT)
- Arm B: RSI predicts dose > 60 Gy (Experimental): Participants will receive treatment with RxRSI guided boost to the primary tumor up to 81Gy (2.7Gy/fraction).
  Interventions: Radiation: Genomically Guided Radiation Therapy (RT)
- Arm C: unable to calculate RSI (Experimental): Participants in will receive standard RT dose of 60Gy in 30 fractions targeting the primary tumor and any involved regional lymph nodes.
  Interventions: Radiation: Genomically Guided Radiation Therapy (RT)

INTERVENTIONS:
Radiation: Genomically Guided Radiation Therapy (RT) — Based on the Radiosensitivity Index (RSI) from testing participants tumor sample, participants will receive either standard dose radiation therapy, which is a strength 60Gy or up to 81Gy strength. Radiation treatment is administered 5 days per week for approximately 6 weeks.

SUMMARY:
The purpose of the study is to determine the feasibility of genomically guided radiation therapy (RT) with concurrent chemotherapy in the management of stage II and III non-small cell lung cancer (NSCLC).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of AJCC Stage 2 or Stage 3 unresectable NSCLC as determined by a multidisciplinary oncology team
* Confirmation of NSCLC with availability of fresh tumor biopsy by tissue biopsy which can include adenocarcinoma, squamous cell, large cell carcinoma, or NSCLC not otherwise specified
* Life expectancy >12 weeks
* Normal renal (creatinine <1.5 × upper limit of normal [ULN]), liver (bilirubin < 1.5 × ULN, transaminases <3.0 × ULN, except in known hepatic disease, wherein may be <5 × ULN) and blood counts (white blood cells ≥2.5, neutrophils ≥1000, platelets ≥50, 000, hemoglobin ≥8)
* ECOG 0-1
* Age ≥ 18 years
* Participants with surgery within 14 days should have recovered from all effects of the surgery and be cleared by their surgeon
* There is no limit on prior systemic or therapies
* Women of childbearing potential and sexually active males must commit to the use of effective contraception while on study
* Ability to sign an informed consent form, which can be signed by a family member or health care proxy. Informed consent must be given before any study related procedures occur.

Exclusion Criteria:

* Current or prior participation in a study of an investigational agent or investigational device within 2 weeks of the first dose of study treatment
* Major surgery or significant traumatic injury that has not been recovered from 14 days before the initiation of study drug
* Women who are pregnant or breastfeeding
* History of allergy or hypersensitivity to any of the study drugs or study drug components
* Concurrent brain metastases or leptomeningeal disease
* History of prior malignancy within 2 years prior to screening, with the exception of those with a negligible risk of metastasis or death (e.g., 5-year OS of > 90%), such as but not limited to, non-melanoma skin carcinoma, ductal carcinoma in situ, or stage I endometriod uterine cancer, and others at the discretion of the PI
* Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [eg, colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc]). The following are exceptions to this criterion:
* • Patients with vitiligo or alopecia
* • Patients with hypothyroidism (eg, following Hashimoto syndrome) stable on hormone replacement
* • Any chronic skin condition that does not require systemic therapy
* • Patients without active disease in the last 5 years may be included but only after consultation with the Principal Investigator
* • Patients with celiac disease controlled by diet alone
* Current or prior use of immunosuppressive medication within 14 days before the first dose of durvalumab. The following are exceptions to this criterion:
* • Intranasal, inhaled, topical steroids, or local steroid injections (eg, intra articular injection)
* • Systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or its equivalent
* • Steroids as premedication for hypersensitivity reactions (eg, CT scan premedication)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2023-05-25 (Actual); Primary Completion 2023-11-29 (Actual); Study Completion 2024-08-21 (Actual)

PRIMARY OUTCOMES:
Rate of Unacceptable Toxicity | 12 weeks after start of treatment
  Rate of Unacceptable Toxicity will be measured during 12 week period following study enrollment. Unacceptable toxicity is defined as any grade 4 or 5 adverse event (AE) probably or definitely related to experimental dose escalated radiation therapy

SECONDARY OUTCOMES:
Freedom from local regional progression (FFLRP) | At 2 years
  Freedom from local regional progression (FFLRP) will be defined as lack of progression as documented by response assessment imaging following completion of concurrent chemotherapy and radiation.
Overall Survival (OS) | At 2 years
  Overall Survival (OS) will be measured from the date of first treatment to the date of death due to any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Dilling, MD, Principal Investigator — Moffitt Cancer Center
Locations (1):
- Moffitt Cancer Center, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: No